CLINICAL TRIAL: NCT05617742
Title: 68Ga-FAPI PET in Evaluation of the Patient With Known or Suspected Lung Cancer: Comparison With Standard 18F-FDG PET
Brief Title: Comparison of 68Ga-FAPI-46 PET and 18F-FDG PET in Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, HO, KUNG-CHU, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202101258A0
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer
Keywords: 68Ga-FAPI-46; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI-46 PET Scan (Experimental): A single-center prospective interventional single-arm clinical trial. All patients will undergo whole-body 68Ga-FAPI-46 PET scan within two weeks before or after 18F-FDG-PET. Injected activity of 68Ga-FAPI-46 is limited to 100-250 MBq per examination.
  Interventions: Diagnostic Test: 68Ga-FAPI-46

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI-46 — 68Ga-FAPI-46 is a radioactive diagnostic agent for PET imaging in the detection of Fibroblast Activation Protein (FAP) positive tumor cells in cancer patients

SUMMARY:
This is a prospective, single-center, single arm, open label study to evaluate the performance of 68Ga-FAPI-46 for the diagnosis of primary and metastatic lesions of lung cancer with comparison to 18F-FDG PET.

DETAILED DESCRIPTION:
FDG-PET imaging is recommended by clinical guidelines for staging of lung cancer; however, there are still limitations of FDG-PET in lung cancer staging due to false-positive and false-negative findings. 68Ga-FAPI PET images have shown high diagnostic performance with high tumor-to-background ratio in various cancers. The purpose of this study is head-to-head comparison of 68Ga-FAPI-46 PET and 18F-FDG PET for the diagnosis and staging or re-staging of lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 20 years
2. Informed consent obtained from patients and families
3. Patients with histology confirmed lung cancer or patients with GGO on chest CT planned to have biopsy or surgery
4. Patients scheduled to undergo FDG-PET examination
5. Performance status: 0, 1, 2, 3

Exclusion Criteria:

1. Contraindication to FAPI-PET and FDG-PET such as pregnant, or lactating patients
2. Patients with mainly malignant pleural effusion without other measurable lesions
3. Undergoing irradiation at accrual
4. Active infection or other serious underlying medical conditions not compatible with study entry
5. History of significant neurological or psychiatric disorders including dementia that would prohibit the understanding and giving of informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To define the diagnostic performance 68Ga-FAPI PET | Through study completion, 2 years
  To evaluate the diagnostic performance (sensitivity, specificity, accuracy) of the 68Ga-FAPI-46 PET scan for identification and staging of lung cancer with comparison to 18F-FDG PET. Histopathology and clinical follow-up will be used as truth standard.

SECONDARY OUTCOMES:
To determine the safety profile of 68Ga-FAPI PET | Up to 7 days post injection with 68Ga-FAPI-46
  Number of participants with 68Ga-FAPI-46 PET scan related adverse events assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Kung-Chu Ho, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Nuclear Medicine, Chang Gung Memorial Hospital, Taoyuan District, Taiwan